CLINICAL TRIAL: NCT05643365
Title: Factors Affecting Timing of Hypothyroidism Following Radioactive Iodine Therapy Patients With Graves Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abdel-Baset Ahmed Ali Alsanory, Resident in nuclear medicine departement (South Egypt Cancer institute), Assiut University
Other Study IDs: Hypothyroidism after RAI
Record Dates: First submitted 2022-11-25; First posted 2022-12-08 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Radioactive Iodine-Induced Hypothyroidism in Graves Disease Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypothyroidism: decreased hormone levels (FT3 < 3.5 pmol/L, FT4 < 11.5 pmol/L, TSH > 4.78 μU/mL) and symptoms of hypothyroidism within 6 months' follow-up.
  Interventions: Radiation: Radioactive Iodine therapy
- Euthyroidism: normal hormone levels (FT3 3.5 to 6.5 pmol/L, FT4 11.5 to 22.7 pmol/L, TSH 0.55 to 4.78 μU/mL), and no symptoms of hyperthyroidism after 6 months' follow-up
  Interventions: Radiation: Radioactive Iodine therapy
- Hyperthyroidism: increased hormone levels (FT3 > 6.5 pmol/L, FT4 > 22.7 pmol/L, TSH < 0.55 μU/mL) and symptoms of hyperthyroidism after 6 months' follow-up
  Interventions: Radiation: Radioactive Iodine therapy

INTERVENTIONS:
Radiation: Radioactive Iodine therapy — All the patient need to stop ATD and iodine-containing drugs for 5 days prior to RAI treatment, and followed a low-iodine diet for 2 weeks. After fasting and water deprivation for 8 h, all the patients took RAI orally in the morning. After taking RAI, the patients need to continue fasting and water deprivation for extra 2 h to avoid the effects of food on iodine absorption.

SUMMARY:
The purpose of this retrospective study was to clarify the possible risk factors of early hypothyroidism after RAI therapy in Graves' disease.

DETAILED DESCRIPTION:
Hyperthyroidism is a clinical syndrome caused by increased thyroid hormone in the blood, it can lead to multiple complications, including cardiac, hepatic, and hematologic system complications. More than 80% of hyperthyroidism are caused by Graves' disease (GD). 3% of women and 0.5% of men may suffer GD in their lifetime [1].

Radioactive iodine (RAI) therapy is an important treatment option for Graves' disease (GD), the main side effect of RAI treatment is hypothyroidism, and the factors resulting in hypothyroidism are still controversial [2]. Male gender, smaller thyroid weight, higher thyroid-stimulating hormone, and smaller thyroid volume are Suggested to be the main risk factors for early hypothyroidism [2]-[3].

ELIGIBILITY:
Inclusion Criteria:

1. Graves' disease patients after one year of RAI therapy .
2. Suppressed serum thyrotropin (TSH) <0.55 µU/ml , elevated serum free triiodothyronine (FT3) > 6.5 pmol/L , free thyroxin FT4 >22.7 pmol/L .

Exclusion Criteria:

1. Patients with other causes of hyperthyroidism , such as toxic multinodular goiter and single toxic adenoma
2. Thyroid cancer
3. Recurrent GD
4. Previous Thyroid surgery
5. Patients can't complete the follow -up within 6 months.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All thyrotoxic patients treated with RAI
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
predictive factors of early hypothyroidism after RAI therapy | 1 year
  Retrospective study from 2013 to 2022 to analyze the correlation between clinical, demographic& and laboratory data and incidence of hypothyroidism by measuring thyroid function tests

SECONDARY OUTCOMES:
the incidence of hypothyroidism within 1 year | 10 years
  To detect the frequency of hypothyroidism after RAI and when it is most likely occur after 6 months or one year

CONTACTS AND LOCATIONS:
Overall Officials: Hemat A Mahmoud, M.D, Study Director — Lecturer; Hanan G Mostafa, M.D, Study Chair — Professor
Locations (1):
- Nuclear medicine unit, department of clinical oncology and nuclear medicine, Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Smith TJ, Hegedus L. Graves' Disease. N Engl J Med. 2016 Oct 20;375(16):1552-1565. doi: 10.1056/NEJMra1510030. No abstract available. PMID 27797318
- [Background] Hu RT, Liu DS, Li B. Predictive factors for early hypothyroidism following the radioactive iodine therapy in Graves' disease patients. BMC Endocr Disord. 2020 May 29;20(1):76. doi: 10.1186/s12902-020-00557-w. PMID 32471411
- [Background] Demir BK, Karakilic E, Saygili ES, Araci N, Ozdemir S. Predictors of Hypothyroidism Following Empirical Dose Radioiodine in Toxic Thyroid Nodules: Real-Life Experience. Endocr Pract. 2022 Aug;28(8):749-753. doi: 10.1016/j.eprac.2022.05.001. Epub 2022 May 7. PMID 35537668